CLINICAL TRIAL: NCT05025839
Title: Long-term Neurological Outcome After SARS-CoV-2 Infection
Brief Title: Neurological Outcome After SARS-CoV-2 Infection
Acronym: ATTRACT
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Medical University Innsbruck (Other)
Responsible Party: Sponsor
Other Study IDs: KLI 986
Record Dates: First submitted 2021-08-18; First posted 2021-08-27 (Actual); Last update posted 2021-08-27 (Actual); Status verified 2021-08

CONDITIONS: SARS-CoV-2; Post-acute COVID-19 Syndrome
MeSH Terms: conditions — Post-Acute COVID-19 Syndrome | interventions — Observation

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (5):
- C healthy: Healthy control group
  Interventions: Other: No Intervention
- C pneum: Control group of patients who were hospitalised and diagnosed with pneumonia ( COVID-19 pneumonia excluded)
  Interventions: Other: No Intervention
- Mild: Outpatients presenting to the hospital with COVID-19
  Interventions: Other: No Intervention
- Moderate: In-patients with COVID-19 not requiring ICU admission
  Interventions: Other: No Intervention
- Severe: Patients with COVID-19 admitted to the ICU
  Interventions: Other: No Intervention

INTERVENTIONS:
Other: No Intervention — No Intervention takes place, Patients are being observed and classified according to disease severity
  Other Names: Observation

SUMMARY:
Wider research context: Since the recognition of SARS-CoV-2 outbreak in 2019, there are now over 126 million COVID-19 cases worldwide with more than 2.7 million deaths. Reports on neurological manifestations vary in prevalence rates (6-84%) and range from mild (headache, hyposmia, myalgia) to severe (encephalopathy, strokes, seizures). Little is known about long-term neurological outcomes of COVID-19 patients. The investigators propose a structured protocol to capture persistent and delayed neurological manifestations, neurocognitive deficits and quality of life (QoL) 3 and 12 months after COVID-19. Objectives: The investigators hypothesize that neurological manifestations and neuropsychological/cognitive deficits can be detected after COVID-19, substantially impact on patients' QoL and can be correlated with structural neuroimaging findings. Main objectives are to assess firstly long-term prevalence rates and natural history of neurological manifestations, secondly neuropsychological/cognitive deficits after COVID-19, thirdly the impact of COVID-19 on measures of mental health, QoL and functional outcome, fourthly to correlate neurological manifestations and distinct neurocognitive deficits with structural MRI abnormalities, and Fifthly to compare these results to age- and sex matched controls hospitalized with pneumonia (Cpneum) and to healthy controls for MRI-data (Chealthy). Approach: The investigators aim to enrol at least 225 patients with COVID-19, in addition to 50 Cpneum and 80 Chealthy. COVID-19 patients will include (group Oóne) outpatients presenting to the hospital, (group two) in-patients not requiring ICU admission, and (group three) patients admitted to the ICU. The investigators will not include asymptomatic patients, patients not presenting to the hospital, and those who do not consent to participate. The standardized protocol includes a firstly a structured neurological examination, secondly olfactory testing, thirdly assessment of QoL, mental health and functional outcome at 3 and 12 months, and fourthly screening for cognitive deficits (at 3 months) and a structured neuropsychological testing (at 12 months) in COVID-19 patients and controls. In a subset of at least 120 COVID-19 patients and 50 controls (Cpneum) high field MRI will be performed at 3 and 12 months. Innovation: The investigators aim to quantify COVID-19 related and specific neurological manifestations and their impact on the individual health condition. The novelty lies in the prospective design, the longitudinal follow-up including and the inclusion of a control group which allows us to explore the natural history of COVID-19 related neurological manifestations. Preliminary analysis of our ongoing 3-month follow-up suggests persistent neurological manifestations and a significant impact of COVID-19 on mental health, cognition and QoL. The investigators believe that our study results likely influence the long-term care of COVID-19 patients and help to identify those, who need further neuro-rehabilitative support

ELIGIBILITY:
Inclusion Criteria:

* (1) Patients of either sex, aged ≥18 years with
* (2) confirmed SARS-CoV-2 infection (according to the Austrian Federal Ministry of Social Affairs, Health, Care and Consumer Protection),
* (3) signed and dated declaration of consent by the patient according to ICH-GCP Guidelines,
* (4) being able to speak and understand the German language

Exclusion Criteria:

* (1) Pre-existing dementia,
* (2) confirmed pregnancy,
* (3) patients without the capacity to consent,
* (4) asymptomatic patients,
* (5) patients not presenting to the hospital

Specific Inclusion/exclusion criteria for the MRI substudy

Inclusion criteria:

* (1) Patients of either sex, aged ≥18 years with
* (2) confirmed SARS-CoV-2 infection (according to the Austrian Federal Ministry of Social Affairs, Health, Care and Consumer Protection),
* (3) signed and dated declaration of consent by the patient according to ICH-GCP Guidelines,
* (4) being able to speak and understand the German language
* (5) agree to participate for MRI

Exclusion criteria:

* (1) Pre-existing dementia,
* (2) confirmed pregnancy,
* (3) patients without the capacity to consent,
* (4) asymptomatic patients,
* (5) patients not presenting to the hospital
* (6) definite contraindication to MRI (e.g. pacemakers)

Controls Patients after pneumonia (Cpneum) We will enrol at least 50 hospitalized age- and sex matched patients with pneumonia based on disease severity during the acute disease as: (group One) hospitalized (moderate; n=25) and (group two) severe patients admitted to the ICU for mechanical ventilation (n=25).

Inclusion criteria:

* (1) Patients of either sex, aged ≥18 years with
* (2) bacterial pneumonia according to CDC criteria,
* (3) signed and dated declaration of consent by the patient according to ICH-GCP Guidelines, and
* (4) being able to speak and understand the German language,
* (5) agree to participate for MRI

Exclusion criteria:

* (1) Pre-existing dementia,
* (2) confirmed pregnancy,
* (3) patients without the capacity to consent,
* (4) definite contraindication to MRI (e.g. pacemakers)

Healthy referents (Chealthy) Currently n=38 MRI acquisitions of prospectively recruited healthy individuals are available, fulfilling the criteria of this proposal (age- and sex matched; same MR protocol). This cohort will be prospectively extended by n=42 to reach age and sex matched criteria.

Ages: 18 Years to 130 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: We aim to include a full dataset of at least 180 patients undergoing 3- and 12-month follow-up. Due to an estimated dropout rate of ~20%, approximately 225 patients are planned to be included in 3-month follow-up. Out of these, we estimate to include a minimum of 50 patients in each of the 3 pre-defined groups, which is feasible based on the preliminary analysis of patient distribution: severe patients: 25%, moderate patients: 50% and mild patients: 25%. In addition, we aim to include at least 120 patients in the MRI sub-study. For the control group, we plan to include 50 age- and sex matched patients (n=25 normal ward, n=25 ICU admission) who undergo the same 3- and 12-month study protocol including MR imaging and neurocognitive testing as COVID-19 patients. Out of these, we expect an estimated dropout rate of ~10% at the 12-month follow-up resulting in 40 patients who will completely finish the study protocol.
Sampling Method: Probability Sample
Enrollment: 355 (Estimated)
Dates: Start 2021-04-07 (Actual); Primary Completion 2023-09-01 (Estimated); Study Completion 2024-09-01 (Estimated)

PRIMARY OUTCOMES:
Prevalence of neurological manifestations in COVID-19 patients | 3-months
  3-month prevalence of neurological manifestations in COVID-19 patients presenting to the hospital in comparison to control patients (Cpneum)
Prevalence of neurological manifestations in COVID-19 patients | 12-months
  12-month prevalence of neurological manifestations in COVID-19 patients presenting to the hospital in comparison to control patients (Cpneum)

SECONDARY OUTCOMES:
Association, prevalence and classification of neurologic manifestations with structural neuroimaging in hospitalised COVID-19 patients after 3-months. | 3-months
  Association of neurologic manifestations (specifically neuropsychological deficits and smelling deficits) with structural neuroimaging (high-field MRI) in comparison to control patients (Cpneum). Prevalence and classification of neuroimaging abnormalities in hospitalized COVID-19 patients in comparison to controls (Cpneum and Chealthy). Other (exploratory) endpoints derived from the clinical database might be analyzed on data driven considerations 3-months after acute disease.
Association, prevalence and classification of neurologic manifestations with structural neuroimaging in hospitalised COVID-19 patients after 12-months. | 12-months
  Association of neurologic manifestations (specifically neuropsychological deficits and smelling deficits) with structural neuroimaging (high-field MRI) in comparison to control patients (Cpneum). Prevalence and classification of neuroimaging abnormalities in hospitalized COVID-19 patients in comparison to controls (Cpneum and Chealthy). Other (exploratory) endpoints derived from the clinical database might be analyzed on data driven considerations 12-months after acute disease.

CONTACTS AND LOCATIONS:
Locations (1):
- Medical University Innsbruck, Department of Neurology, Innsbruck, Tyrol, Austria

IPD SHARING:
Plan to Share IPD: No